CLINICAL TRIAL: NCT00266669
Title: Phase III "in-Life" Study of a Topical Gel Formulation of Nitroglycerin, MQX-503, and Matching Placebo Gel in the Treatment and Prevention of Raynaud's Phenomenon
Brief Title: Phase III Study of Topical Gel for Treatment and Prevention of Raynaud's Phenomenon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MediQuest Therapeutics (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 05-002; MQX-503 In-Life
Record Dates: First submitted 2005-12-15; First posted 2005-12-19 (Estimated); Last update posted 2007-08-08 (Estimated); Status verified 2007-08

CONDITIONS: Raynaud's Disease
Keywords: Raynaud's Phenomenon; Raynaud's Disease; Scleroderma; Raynaud's Disease Secondary to Scleroderma; Raynaud's Disease Secondary to Other Autoimmune Disease
MeSH Terms: conditions — Raynaud Disease; Scleroderma, Diffuse | interventions — Nitroglycerin

INTERVENTIONS:
Drug: Topical organogel with nitroglycerin

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of a topical gel formulation of nitroglycerin, in comparison to a matching placebo, for patients with moderate to severe primary Raynaud's phenomenon or patients with Raynaud's phenomenon secondary to autoimmune diseases, such as scleroderma.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Raynaud's phenomenon
* 2 or more Raynaud's events on a typical winter day
* Agree to discontinue current treatments for Raynaud's
* Negative pregnancy test and agree to use effective contraception during study

Exclusion Criteria:

* Current use of nitrate medications or medications known to interact with nitroglycerin
* Patients who currently use medications, like calcium channel blockers, that might interfere with study medication
* Patients with a known allergy to nitroglycerin or common topical ingredients
* Patients with a history of migraine headaches
* Patients with a history of unstable medical problems
* Patients with cognitive or language difficulties that would impair completion of assessment instruments
* Patients with lab screening values more than 20% outside normal range
* Patients with non-epithelialized skin lesions, in the area where the gel is to be applied, at the time of screening
* Pregnant or nursing women
* Women of child-bearing potential who are unwilling to comply with the contraceptive requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2005-12; Study Completion 2006-05

PRIMARY OUTCOMES:
Improvements in Raynaud's Assessment Score comparing active to placebo
Reduction of number of Raynaud's events
Decrease in duration of Raynaud's events
Decrease in symptoms associated with Raynaud's
Assess safety: frequency and severity of adverse events associated with the study drug

SECONDARY OUTCOMES:
Improvement in patient's health using physician's Global Assessment and patient's Heath Assessment Questions
Reduction in emergence of digital ulcers for patients with scleroderma

CONTACTS AND LOCATIONS:
Locations (19):
- United States (17):
  - Stanford Medical School, Stanford, California
  - University of Colorado at Denver and Health Sciences Center, Denver, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Center for Advanced Medicine, Chicago, Illinois
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Arthritis Education & Treatment Center, PLLC, Grand Rapids, Michigan
  - University of Medicine and Dentistry of New Jersey, New Brunswick, New Jersey
  - The Center for Rheumatology, Albany, New York
  - SUNY Stony Brook, East Setauket, New York
  - Duke University, Durham, North Carolina
  - Medical University of Ohio, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Medical School at Houston, Houston, Texas
  - Virginia Mason Benaroya Research Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - St. Joseph's Health Care, London, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec